CLINICAL TRIAL: NCT01249118
Title: A Phase 1, Single Dose, Randomized, Cross-over Absolute Bioavailability Study in Healthy Subjects Comparing Oral to Intravenous Administration of GDC-0973
Brief Title: An Absolute Bioavailability Study in Healthy Participants Comparing Oral to Intravenous Administration of GDC-0973 (Cobimetinib)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MEK4952g
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — cobimetinib

ARMS (3):
- Part 1: GDC-0973 IV Infusion First, Then GDC-0973 Capsules (Experimental): Participants will receive single dose of GDC-0973 2 milligrams (mg) IV infusion in first intervention period followed by single dose of GDC-0973 20 mg oral capsules (four 5-mg capsules) in second intervention period. The washout period between each period will be a minimum of 10 days.
  Interventions: Drug: GDC-0973 IV Infusion; Drug: GDC-0973 Oral Capsules
- Part 2: GDC-0973 IV Infusion First, Then GDC-0973 Capsules (Experimental): Participants will receive single dose of GDC-0973 2 mg IV infusion in first intervention period followed by single dose of GDC-0973 20 mg oral capsules (four 5-mg capsules) in second intervention period. The washout period between each period will be a minimum of 10 days.
  Interventions: Drug: GDC-0973 IV Infusion; Drug: GDC-0973 Oral Capsules
- Part 2: GDC-0973 Capsules First, Then GDC-0973 IV Infusion (Experimental): Participants will receive single dose of GDC-0973 20 mg oral capsules (four 5-mg capsules) in first intervention period followed by single dose of GDC-0973 2 mg IV infusion in second intervention period. The washout period between each period will be a minimum of 10 days.
  Interventions: Drug: GDC-0973 IV Infusion; Drug: GDC-0973 Oral Capsules

INTERVENTIONS:
Drug: GDC-0973 IV Infusion — IV infusion.
  Other Names: XL518
Drug: GDC-0973 Oral Capsules — Oral dose.
  Other Names: XL518

SUMMARY:
The primary objective of Part 1 of this study is to evaluate the safety and tolerability of the intravenous (IV) dose of GDC-0973. The primary objectives of Part 2 of this study are to evaluate the absolute bioavailability of GDC-0973 and to evaluate the pharmacokinetic (PK) of GDC-0973 following IV and oral administration. The secondary objective of Part 2 of this study is to evaluate the safety of GDC-0973 administered orally and intravenously.

ELIGIBILITY:
Inclusion Criteria

* Within body mass index range 18.5 to 29.9 kilograms per square meter (kg/m^2)
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiogram (ECG), and vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory
* Negative test for selected drugs of abuse at Screening and at each Check-in
* Negative hepatitis panel and anti-hepatitis C virus and negative human immunodeficiency virus (HIV) antibody screens
* Healthy males and females of non-child-bearing potential or who agree to use effective contraception

Exclusion Criteria

* Significant history or clinical manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy, hernia repair, and cholecystectomy will be allowed
* History or presence of an abnormal ECG
* History of alcoholism or drug addiction prior to period 1 check-in
* Use of any tobacco-containing or nicotine-containing products prior to period 1 check-in
* Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 28 days or 5 half-lives, whichever is longer, prior to period 1 check-in
* Use of any prescription medications/products, including proton pump inhibitors, within 14 days prior to period 1 check-in
* Poor peripheral venous access
* Any acute or chronic condition that would limit the participants ability to complete and/or participate in this clinical study
* Female participant is pregnant, lactating, or breastfeeding
* Predisposing factors to retinal vein occlusion (RVO)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Rooney, M.D., PhD, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was divided into two parts. In part 1 of the study, safety of GDC-0973 was evaluated and in part 2 pharmacokinetics (PK) of GDC-0973 was evaluated. All PK outcomes apply only to part 2 of the study while safety applies to part 1 and 2 both.
Groups:
- Part 1: GDC-0973 IV Infusion First, Then GDC-0973 Capsules: Participants received single dose of GDC-0973 2 milligrams (mg) intravenous (IV) infusion in first intervention period followed by single dose of GDC-0973 20 mg oral capsules (four 5-mg capsules) in second intervention period. There was a washout period of minimum 10 days after each intervention period.
- Part 2: GDC-0973 IV Infusion First, Then GDC-0973 Capsules: Participants received single dose of GDC-0973 2 mg IV infusion in first intervention period followed by single dose of GDC-0973 20 mg oral capsules (four 5-mg capsules) in second intervention period. There was a washout period of minimum 10 days after each intervention period.
- Part 2: GDC-0973 Capsules First, Then GDC-0973 IV Infusion: Participants received single dose of GDC-0973 20 mg oral capsules (four 5-mg capsules) in first intervention period followed by single dose of GDC-0973 2 mg IV infusion in second intervention period. There was a washout period of minimum 10 days after each intervention period.
Period: First Intervention Period
Arm/Group | Part 1: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 Capsules First, Then GDC-0973 IV Infusion
Started | 2 | 6 | 5
Completed | 2 | 6 | 5
Not Completed | 0 | 0 | 0
Period: First Washout Period
Arm/Group | Part 1: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 Capsules First, Then GDC-0973 IV Infusion
Started | 2 | 6 | 5
Completed | 2 | 5 | 5
Not Completed | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Second Intervention Period
Arm/Group | Part 1: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 Capsules First, Then GDC-0973 IV Infusion
Started | 2 | 5 | 5
Completed | 2 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Second Washout Period
Arm/Group | Part 1: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 IV Infusion First, Then GDC-0973 Capsules | Part 2: GDC-0973 Capsules First, Then GDC-0973 IV Infusion
Started | 2 | 5 | 5
Completed | 2 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received study drug and had at least 1 post-dose safety assessment for Part 1 and the participants who were randomized, received study drug, and had at least 1 post-dose safety assessment for Part 2.
Groups:
- Entire Study Population: Part 1: Participants received single dose of GDC-0973 2 mg IV infusion in first intervention period followed by single dose of GDC-0973 20 mg oral capsules (four 5-mg capsules) in second intervention period. There was a washout period of minimum 10 days after each intervention period.
  Part 2: Participants received single dose of GDC-0973 2 mg IV infusion and GDC-0973 20 mg oral capsules (four 5-mg capsules) in either of the two intervention periods. There was a washout period of minimum 10 days after each intervention period.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of IV and Oral GDC-0973
Time Frame: Part 2: 0 hours (Hrs) (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population included participants who were randomized, received study drug, and had at least 1 valid PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- GDC-0973 2 mg IV: Participants received single dose of GDC-0973 2 mg IV infusion in either of the intervention periods in part 2 of the study.
- GDC-0973 20 mg Oral: Participants received single dose of GDC-0973 20 mg oral capsules (four 5-mg capsule) in either of the intervention periods in part 2 of the study.
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
nanograms per milliliter (ng/mL) | 20.5 (35.6) | 15.2 (26.4)

2. Primary Outcome: Dose Normalized Cmax [Cmax(dn)] of IV and Oral GDC-0973
Description: Cmax(dn) is Cmax divided by dose.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
ng/mL/mg | 10.2 (35.6) | 0.844 (26.4)
Statistical Analysis 1: Comparison: GDC-0973 2 mg IV vs GDC-0973 20 mg Oral; Least squares (LS) mean was calculated from analysis of variance (ANOVA). Data for dose-normalized Cmax were natural log-transformed prior to analysis; Test type: Superiority or Other; Ratio of LS Means = 8.45, 90% CI 2-sided [7.08 to 10.08] — The 90 percent (%) confidence intervals (CI) of test group (oral dose) means relative to reference group (IV dose) means were obtained by taking antilog of corresponding 90% CI for the differences between the means on the log scale

3. Primary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of IV and Oral GDC-0973
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
ng/mL | 0.261 (37.1) | 0.546 (70.0)

4. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of IV and Oral GDC-0973
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Median (Full Range); unit: hr
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
hr | 0.500 [0.500 to 0.567] | 4.00 [2.00 to 8.00]

5. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of IV and Oral GDC-0973
Description: AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t).
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
ng*hr/mL | 156 (19.1) | 688 (28.4)

6. Primary Outcome: Dose Normalized AUC (0-t) [AUC (0-t)dn] of IV and Oral GDC-0973
Description: AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t). AUC (0-t)dn is AUC (0-t) divided by dose.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
ng*hr/mL/mg | 77.8 (19.1) | 38.2 (28.4)
Statistical Analysis 1: Comparison: GDC-0973 2 mg IV vs GDC-0973 20 mg Oral; LS means was calculated from ANOVA. Data for dose-normalized AUC (0 - t) were natural log-transformed prior to analysis; Test type: Superiority or Other; Ratio of LS Means = 48.6, 90% CI 2-sided [41.43 to 56.94] — The 90% CI of the test group (oral dose) means relative to the reference group (IV dose) means were obtained by taking the antilog of the corresponding 90% CI for the differences between the means on the log scale

7. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of IV and Oral GDC-0973
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
ng*hr/mL | 188 (16.2) | 784 (29.5)

8. Primary Outcome: Dose Normalized AUC (0 - ∞) [AUC (0 - ∞)dn] of IV and Oral GDC-0973
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). AUC (0 - ∞)dn is AUC(0 - ∞) divided by dose.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL/mg
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
ng*hr/mL/mg | 93.9 (16.2) | 43.5 (29.5)
Statistical Analysis 1: Comparison: GDC-0973 2 mg IV vs GDC-0973 20 mg Oral; LS mean was calculated from ANOVA. Data for dose-normalized AUC (0 - ∞) were natural log-transformed prior to analysis; Test type: Superiority or Other; Ratio of LS Means = 45.9, 90% CI 2-sided [39.74 to 53.06] — [estimate comment as in outcome 6, analysis 1]

9. Primary Outcome: Plasma Decay Half-Life (t1/2) of IV and Oral GDC-0973
Description: t1/2 is the time measured for the plasma concentration of GDC-0973 to decrease by one half.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
hr | 73.8 (17.1) | 66.2 (18.2)

10. Primary Outcome: Systemic Clearance (CL) of IV GDC-0973
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population who received IV dose of GDC-0973.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)/hr
Arm/Group | GDC-0973 2 mg IV
Number analyzed (Participants) | 11
Liter (L)/hr | 10.7 (16.2)

11. Primary Outcome: Apparent Oral Clearance (CL/F) of Oral GDC-0973
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modelling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population who received oral dose of GDC-0973.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | GDC-0973 20 mg Oral
Number analyzed (Participants) | 10
L/hr | 23.0 (29.5)

12. Primary Outcome: Volume of Distribution at Steady State (Vss) of IV GDC-0973
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose of Day 1
Population: Full analysis population who received IV dose of GDC-0973.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | GDC-0973 2 mg IV
Number analyzed (Participants) | 11
Liter | 1052 (28.2)

13. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Oral GDC-0973
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/F is influenced by the fraction absorbed.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population who received oral dose of GDC-0973.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | GDC-0973 20 mg Oral
Number analyzed (Participants) | 10
Liter | 2197 (31.9)

14. Primary Outcome: Absolute Oral Bioavailability (F) of GDC-0973
Description: Absolute oral bioavailability is the amount of drug from a formulation that reaches the systemic circulation relative to an IV dose. F = [AUC (0-∞), oral multiplied by Dose IV] divided by [AUC (0-∞), IV multiplied by Dose oral]. Absolute oral bioavailability is determined for drugs which are administered orally. IV dose is 100% in systemic circulation (dosed directly) and hence no estimation is required.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population who received oral dose of GDC-0973.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | GDC-0973 20 mg Oral
Number analyzed (Participants) | 10
Ratio | 0.457 (25.0)

15. Primary Outcome: Mean Absorption Time (MAT)
Description: MAT is mean time required for the drug to reach the central compartment. MAT was estimated from the mean resident time (MRT) from oral and IV administration. MAT was calculated as MRT last of oral dose minus MRT last of IV dose. MAT is analyzed when drug is administered orally (only for non-IV routes of administration).
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1
Population: Full analysis population who received oral dose of GDC-0973. Here, "number of participants analyzed" signified those participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | GDC-0973 20 mg Oral
Number analyzed (Participants) | 4
hr | 2.67 (58.0)

16. Primary Outcome: Amount of Drug Excreted in the Urine (Aeu) of IV and Oral GDC-0973
Description: The cumulative amount of drug excreted in urine over the entire collection interval of 96 hrs was calculated by adding the Aeu of the intervals 0 to 12, 12 to 24, 24 to 48, 48 to 72, and 72 to 96 hrs where Aeu was calculated by multiplying the urine volume within the collection interval by the associated drug concentration.
Time Frame: Part 2: 0 to 12, 12 to 24, 24 to 48, 48 to 72, and 72 to 96 Hrs post-dose on Day 1
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
mg | 0.0761 (22.3) | 0.379 (33.9)

17. Primary Outcome: Renal Clearance (CLR) of IV and Oral GDC-0973
Description: CLR was calculated as Aeu divided by AUC (0 - ∞), where Aeu was amount of drug excreted in urine from time 0 to 96 hrs post-dose and AUC(0 - ∞) was area under the concentration-time curve of the analyte in plasma over the time interval from zero extrapolated to infinity hrs post-dose.
Time Frame: Part 2: 0 Hrs (pre-dose), 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 144, and 192 Hrs post-dose on Day 1 for plasma; 0 to 12, 12 to 24, 24 to 48, 48 to 72, and 72 to 96 Hrs post-dose for urine
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
L/hr | 0.405 (20.1) | 0.484 (22.4)

18. Primary Outcome: Percent of GDC-0973 Excreted in the Urine (% Excreted) for IV and Oral GDC-0973
Description: % Excreted is the mean percentage of dose recovery in urine and calculated as: (Aeu divided by dose) multiplied by 100, where Aeu was amount of drug excreted in urine from time 0 to 96 hrs post-dose.
Time Frame: Part 2: 0 to 12, 12 to 24, 24 to 48, 48 to 72, and 72 to 96 Hrs post-dose
Population: Full analysis population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percent dose excreted
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Number analyzed (Participants) | 11 | 10
Percent dose excreted | 3.81 (22.3) | 1.90 (33.9)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from start of study treatment in first period to end of second period (up to 30 days)
Description: Safety population. One participant discontinued study in first period (Part 2) and did not receive GDC-0973 20 mg oral dose in second period. Therefore, only 12 participants were evaluable for adverse events in this treatment arm.
Groups:
- GDC-0973 2 mg IV: Participants received GDC-0973 2 mg IV infusion in either intervention period in part 1 and part 2 of the study.
- GDC-0973 20 mg Oral: Participants received GDC-0973 20 mg oral capsules (four 5-mg capsule) in either intervention period in part 1 and part 2 of the study.
Arm/Group | GDC-0973 2 mg IV | GDC-0973 20 mg Oral
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 2/13 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GDC-0973 2 mg IV (N=13) | GDC-0973 20 mg Oral (N=12)
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Feeling hot (General disorders) | 0 | 1
Infusion site erythema (General disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.